CLINICAL TRIAL: NCT06591533
Title: The Effect of Music Therapy on Vital Signs and Heart Rate Variability of Pediatric Patients During the Extubation Process in the Pediatric Intensive Care Unit
Brief Title: The Effect of Music Therapy on Vital Signs and Heart Rate Variability of Pediatric Patients During the Extubation Process.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Claudia Aristizábal (Other)
Collaborators: Sanitas University (Other)
Responsible Party: Sponsor-Investigator, Claudia Aristizábal, Director, Sanitas University
Organization: Sanitas University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: INV-MT EXTUBACION
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Respiratory Failure; Intensive Care Pediatric
Keywords: vital signs; Pediatric Intensive Care Unit; extubation; music therapy; mechanical ventilation; hear rate
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Music Therapy; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Music therapy + standard care (Experimental)
  Interventions: Other: Music therapy + standard care
- Standard care (Other)
  Interventions: Other: Standard Care (in control arm)

INTERVENTIONS:
Other: Music therapy + standard care — In the pre-extubation and extubation phase, the musical characteristics will be based on a slow to medium tempo, simple harmonic structures (e.g., tonic-subdominant movements), fluid melodies, and avoiding large intervals or abrupt changes of tonalities. The musical instruments used will be a classical guitar with nylon strings (Yamaha C-40) and the voice of the music therapist without lyrics or words. In the post-extubation phase, the musical characteristics will be based on a moderate tempo, introducing chord progressions aiming at tension-resolution (e.g., dominant-tonic), and a more rhythmic application of melodic or harmonic material.
  Arms: Music therapy + standard care
Other: Standard Care (in control arm) — Standard care during the extubation process involves providing usual the medical care provided for patients according to each hospital's guidelines.
  Arms: Standard care

SUMMARY:
The extubation process is critical to the future health outcomes of the pediatric patient because it tests the ability of the respiratory system to function without the support of mechanical ventilation. However, extubation can cause stress, pain, anxiety, or discomfort in the patients, which results in an increased likelihood of reintubation. Music therapy has been shown to be effective in reducing anxiety and stress levels in ventilated adult patients, but studies evaluating the effect of music therapy on vital signs in pediatric patients during extubation are lacking.

The aim is to determine the effect of music therapy on vital signs and heart rate variability of pediatric patients during extubation in in two high-complexity health care institutions in Colombia.

This study is a Randomized clinical trial (RCT) with two parallel arms. The intervention group (IG) will receive standard care during the extubation process + music therapy and the control group (CG) will receive standard care only. The primary outcome measure is heart rate (HR) measured every minute for 5 minutes before extubation, during extubation, and up to 10 minutes after extubation. Secondary measures are: oxygen saturation, respiratory rate, blood pressure, duration of the procedure, number of reintubations, and heart rate variability.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients hospitalized who are undergoing an extubation process.

Exclusion Criteria:

* Pediatric patients with accidental extubation will be excluded.

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 82 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Heart rate | From 5 minutes pre-extubation to 10 minutes post-extubation.
  It will be measured through pulse oximetry every minute.

SECONDARY OUTCOMES:
Respiratory rate | From 5 minutes pre-extubation to 10 minutes post-extubation.
  It will be measured through pulse oximetry every minute.
Oxygen saturation | From 5 minutes pre-extubation to 10 minutes post-extubation.
  It will be measured through pulse oximetry every minute.
Blood pressure | From 5 minutes pre-extubation to 10 minutes post-extubation.
  Diastolic, systolic, and mean BP will be measured on the forearm with an age-appropriate cuff, at the level of the brachial artery in the right antecubital fossa, every 5 minutes.
Heart rate variability | From 5 minutes pre-extubation to 10 minutes post-extubation.
  It will be measured with the electrocardiogram by standard monitoring.

CONTACTS AND LOCATIONS:
Locations (2):
- Colombia (2):
  - Clínica Reina Sofia Pediátrica y Mujer, Bogotá, Bogota D.C.
  - Clínica Infantil Santa María del Lago, Bogotá, Bogota D.C.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beltran YM, Charum DP, Zuluaga CA, Vega MA, Benavides-Cruz J, Amarillo M, Canon E, Alvarez I, Ramirez-Moreno J, Paez L, Garzon MC, Calderon PD, Quintero TC, Moreno J, Ettenberger M. Effect of music therapy on vital signs and heart rate variability of paediatric patients during the extubation process in the paediatric intensive care unit: a multicentre randomised clinical trial protocol. BMJ Open. 2025 Nov 19;15(11):e098251. doi: 10.1136/bmjopen-2024-098251. PMID 41263836